CLINICAL TRIAL: NCT06103279
Title: Evaluation of Empagliflozin Effect Against Doxorubicin Induced Cardiomyopathy
Brief Title: Cardioprotective Empagliflozin for Cancer Patients Receiving Doxorubicin
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Abdelrahman Ahmed Abdelsalam Attia, Teaching assistant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Cardioprotective Empagliflozin
Record Dates: First submitted 2023-10-22; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Cancer
Keywords: Empagliflozin; Doxorubicin OR Adriamycin; Cardiomyopathy OR Cardiotoxicity
MeSH Terms: conditions — Neoplasms | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: The work is a prospective, randomized, controlled study. A total of 40 cancer patients who will receive DOX-based chemotherapy will be enrolled in the study
  These patients will be randomly assigned to either Group I or Group II (each group contains 20 patients) Group I: will receive the standard chemotherapy protocol (DOX-based chemotherapy) only.
  Group II: will receive the standard chemotherapy protocol (DOX-based chemotherapy) plus Empagliflozin.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empa Arm (Experimental): (Intervention group = 20 patients) >> will receive the standard chemotherapy protocol (DOX-based chemotherapy) plus Empagliflozin.
  Empagliflozin dose and duration:
  According to the Evidence-based doses of disease-modifying drugs in key randomized trials in patients with heart failure with reduced ejection fraction with or without diabetes, The recommended dose of empagliflozin is 10 mg once daily.
  1 tablet once daily of continuously starting from 1 week before starting DOX till the end of last Dox-based chemotherapy dose according to the given chemotherapy protocol.
  Interventions: Drug: Empagliflozin 10 MG
- Control Arm (No Intervention): (Control group = 20 patients) >> will receive the standard chemotherapy protocol (DOX-based chemotherapy) only.

INTERVENTIONS:
Drug: Empagliflozin 10 MG — 1 tablet once daily of (EMPAGLIMAX® 10 mg) continuously starting from 1 week before starting doxorubicin till the end of last Dox-based chemotherapy dose according to the given chemotherapy protocol
  Arms: Empa Arm

SUMMARY:
Doxorubicin induced cardiomyopathy is the most common and serious side effect associated with doxorubicin treatment in cancer patients receiving doxorubicin. Studies have been shown that Empagliflozin can reduce cardiovascular mortality and hospitalization for heart failure in patients with heart failure with or without diabetes and current clinical trials indicate that SGLT2 inhibitors protect against heart failure outcomes and can reduce cardiac remodeling even in patients without diabetes. Empagliflozin had beneficial effects on the outcome of the cardiomyopathy and also has anti-tumor activity in animal studies, but clinical studies are still lacking. We are going to investigate the cardioprotective effect of Empagliflozin against doxorubicin induced cardiomyopathy.

Objective:

* Evaluate the prophylactic effect of using Empagliflozin "a selective inhibitor of the sodium glucose co-transporter 2 (SGLT2)" against doxorubicin induced cardiotoxicity in patients receiving doxorubicin-based chemotherapy.
* Monitor the safety of adding empagliflozin to doxorubicin-based chemotherapy.

DETAILED DESCRIPTION:
In cancer therapy, several cytotoxic drugs may cause cardiotoxicity which is associated with poor short- and long-term outcome. Anthracyclines (ANT) are natural products with topoisomerase-interacting activity. These compounds are broadly utilized in the treatment of lymphoma, sarcoma, breast cancer, and pediatric leukemia. ANT has long been demonstrated to improve survival in cancer patients. However, despite its broad effectiveness, ANT therapy is associated with irreversible dilated cardiomyopathy (CMP). Toxic effect may occur at any stage of ANT treatment. and it seems that females are affected more often than males. The incidence increases from 5% in patients receiving doses up to 400 mg/m2 to 48% in patients receiving more than 700 mg/m2 of doxorubicin (DOX). Although the risk of cardiac dysfunction is proportional to the cumulative ANT exposure, a substantial number of patients still develop severe cardiotoxicity at doses well below 550 mg/m2. In a study on the early detection and prediction of cardiotoxicity, 27.6% of patients developed chemotherapy-related cardiotoxicity. Another study found that DOX in doses of less than 300 mg/m2 could induce cardiotoxicity. Strategies that might prevent chemotherapy-induced CMP are receiving increased attention from oncologists and cardiologists. It is also well known that most doxorubicin-induced cardiotoxicity occurs within the first year (mainly within 6-months after chemotherapy). Acute toxicity is a reversible adverse effect that develops during or within days of ANT infusion, and its incidence has been significantly reduced by slowing the ANT infusion rates. Congestive heart failure due to chronic cardiotoxicity is the most common type of ANT damage, is irreversible, and peaks at 1-3 months but can occur even years after therapy. Free radical formation is generally accepted as the main mechanism. cardiomyocytes have poor antioxidant defense systems, and free oxygen radicals can damage various targets in the cell. This may result in impairment of cardiac contractility and the development of CMP. Compared with other more common forms of CMP, myocardial damage has been accompanied by a grave prognosis, has a 2-year mortality rate of up to 6 %, and seems to be refractory to therapy. The various approaches that can be employed in clinical practice include dosage restriction; encapsulating ANT in liposomes to reduce myocardial uptake; and simultaneous administration with iron chelator dexrazoxane to reduce the free iron-catalyzed reactive oxygen formation and the alteration of ANT configuration.

Nonetheless, ANT-induced heart failure has morbidity and mortality sequelae. The second evident problem of using DOX as a chemotherapeutic agent is the acquired tumor resistance against it "Multidrug resistance (MDR)". DOX drug resistance is developed as a result of increased expression of the ATP-dependent efflux pump ABCB1 (MDR1), which encodes the membrane drug transporter P-glycoprotein.

Empagliflozin (EMPA) exerts an antidiabetic effect by reducing glucose reabsorption from the renal proximal tubules using sodium-glucose cotransporter-2 (SGLT-2) inhibition. Dissecting the exact molecular mechanism of SGLT2 inhibitors is therefore hampered by the diabetic scenario. Moreover, current clinical trials indicate that SGLT2 inhibitors protect against heart failure outcomes even in patients without diabetes. Beyond its antidiabetic effects, it has been shown to reduce all-cause death, cardiovascular death, and hospitalizations due to heart failure in diabetic patients compared to placebo in the EMPA-REG OUTCOME clinical study. As well, EMPORER reduced clinical trial revealed EMPA reduced cardiovascular mortality and hospitalization for heart failure in patients with heart failure with or without diabetes. The SGLT2 inhibitors canagliflozin, dapagliflozin, empagliflozin, ertugliflozin and sotagliflozin were studied in patients with established CV disease in the EMPAREG OUTCOME and VERTIS-CV trials, with established CV disease or CV risk factors in the CANVAS and DECLARE-TIMI 58 trials, and with CKD and CV risk in the SCORED trial, respectively. EMPA and canagliflozin reduced the primary composite endpoint of major CV adverse events, including CV death or nonfatal MI or non-fatal stroke, and HF hospitalizations in EMPA-REG OUTCOME and CANVAS, respectively. EMPA also reduced all-cause death or CV death alone. The effects on the primary endpoint were driven by the reduction in HF-related events. Many different chemical agents have been examined to prevent ANT-induced CMP and some of them showed promising results. Recent animal studies and experimental observations showed that EMPA prevented the development of CMP, free radical release, and apoptosis in cardiomyocytes due to chemotherapeutics including; DOX. These cardiovascular outcome trials of SGLT2 inhibitors have led to numerous speculations and studies related to their potential protective mechanisms in patients with heart failure. Some of the proposed mechanisms are hemodynamic-related, including natriuresis, osmotic diuresis, blood pressure-lowering, and LV remodeling. Other mechanisms are related to more systemic effects, including the regulation of myocardial energetics, inhibition of sodium-hydrogen exchange, adipokines and myokines, uric acid homeostasis, elevation in erythropoietin levels, increases in endothelial progenitor cells, protection from DOX, and the regulation of autophagy. Despite this, little is currently known about the molecular mechanisms underlying the cardiac protection provided by SGLT2 inhibitors. According to ESC guidelines in Aug.2021, Dapagliflozin or EMPA is recommended for patients with chronic Heart failure with reduced ejection fraction (HFrEF) with or without diabetes to reduce the risk of HF hospitalization and death.

Evidence Class Ia Level Ab. The sodium-glucose co-transporter 2 (SGLT2) inhibitors dapagliflozin and EMPA added to therapy with ACE-I/ARNI/betablocker/MRA reduced the risk of CV death and worsening HF in patients with HFrEF. Unless contraindicated or not tolerated, dapagliflozin or EMPA are recommended for all patients with HFrEF already treated with an ACE-I/ARNI (angiotensin-converting enzyme inhibitor/ angiotensin receptor neprilysin inhibitor), a beta-blocker, and an MRA (mineralocorticoid receptor antagonist), regardless of whether they have diabetes or not. The SGLT2 inhibitor, EMPA, protects the heart from DOX associated CMP in mice, by acting through a novel Beclin 1-toll-like receptor (TLR) 9-sirtuin-(SIRT) 3 axis. EMPA increases the abundance of mitochondrial SIRT3. Also; it enhances the activation of TLR9 to bind with Beclin 1, triggering communication to the autophagic, immune system, and Inflammatory machinery. Further studies also showed that EMPA can protect DOX-induced heart failure in mice. This evidence clearly indicates that SGLT2 inhibitors have direct cardiac protection mechanisms other than glucose modulation. EMPA attenuates the cardiotoxic effects exerted by DOX on LV function and remodeling in nondiabetic mice, independently of glycemic control. EMPA prevents the reduction in cardiac systolic function induced by a cardiotoxic ANT in a model of non-diabetic mice. The protective impact of EMPA on systolic function was also associated with better systolic and diastolic blood pressures in mice treated with EMPA compared to those treated with DOX alone. Finally, histological examination showed a lower degree of myocardial fibrosis in mice treated with EMPA. Also the protective effect of EMPA against DOX cardiotoxicity can be explained by several mechanisms including;

1. EMPA upregulates mitochondrial PGC-1α, thereby increasing mitochondrial biogenesis and protecting mitochondria.
2. EMPA prevents cardiomyocyte apoptosis by reducing sarcoplasmic reticulum degeneration in a significant manner.

4- Prevents the deterioration of left ventricular systolic functions in echocardiography. 5- EMPA markedly attenuates DOX -induced prolongation of the QT and QTc intervals on the ECG through decreasing the amount of cytosolic calcium and decreasing late sodium channel activation in this way can shorten QT interval. 6- Oh et al. showed EMPA improved fractional shortening (FS) but not ejection fraction (EF) in MRI and reduced perivascular and interstitial fibrosis in histologic examination in DOX-induced chronic cardiotoxicity. 7- Protective effects of EMPA on cardiomyocytes originate from an increase in beta-hydroxybutyrate (βoh) (as an antioxidant) level. 8- Decrease in preload and afterload due to natriuresis or the antioxidant effect provided by the elevated levels of antioxidant βoh. EMPA exerts anti-inflammatory and cardioprotective effects in DOXO-induced cardiotoxicity as EMPA inhibits the activity of SGLT-2 thereby reducing intracellular glucose and sodium in cardiomyocytes, resulting in the inhibition of iROS, lipid peroxidation and NLRP3/MyD88-related pathways; the inhibition of NLRP3 and NF-kB reduces the pro-inflammatory cytokine storm in cardiomyocytes exposed to DOXO. Finally, EMPA has shown antitumor activity in different murine cancer models The anti-hyperglycemic drug, EMPA, was recently indicated to have in vitro anticancer potential together with its previously reported cardioprotective properties related to calmodulin inhibition.

* Recently, it was indicated that EMPA has an in vitro anticancer potential against both breast cancer cell lines MCF-7 and lung cancer cell lines (A549.21).
* EMPA has shown cardioprotective properties due to its role as an inhibitor of calmodulin.
* Calmodulin is a calcium-binding protein which is regulating many of the intracellular actions of calcium. It is proposed that calmodulin is responsible for the regulation of cellular proliferation and that its function may be altered in malignancy.
* Mustroph et al. proposed that EMP reduces Ca2+/calmodulin-dependent kinase (CaMKII) activity in isolated murine ventricular myocytes. Also, the diastolic function of heart failure was improved in a nondiabetic rodent model by using EMPA.
* Also; calmodulin antagonists are cytotoxic and can restore the sensitivity of resistant cells to drugs such as DOX and vincristine. Consequently, calmodulin has been suggested as an emerging target for anticancer therapeutic intervention.

The aim of this study is to:

* Evaluate the prophylactic effect of using Empagliflozin "a selective inhibitor of the sodium glucose co-transporter 2 (SGLT2)" against doxorubicin induced cardiotoxicity in patients receiving doxorubicin-based chemotherapy.
* Monitor the safety of adding empagliflozin to doxorubicin-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Chemo-naive patients with a first diagnosis of cancer and indication for first-line therapy with doxorubicin-based chemotherapy.
2. Patients intended to receive at least 4 cycles of doxorubicin or greater.
3. No previous cardiac conditions (including ischemic heart disease and clinically important congenital or acquired valvular and myocardial diseases) and taking no cardiac-related drugs.
4. An echocardiographic LVEF value ≥55%.
5. Normal hepatic and renal function (bilirubin ≤1.5 mg/dL, creatinine ≤2.0 mg/dL).
6. ECOG performance grade 0, 1 or 2.

Exclusion Criteria:

1. Hypersensitivity / Allergy to Empagliflozin.
2. Any condition that contraindicates chemotherapy (i.e., pregnancy, lactation).
3. New-onset cardiac symptoms or presence of congestive heart failure symptoms or established (dilated, restrictive or hypertrophic) cardiomyopathy, coronary heart disease, moderate or severe aortic and/or mitral valve disease or atrial fibrillation detected by baseline echocardiography.
4. Systemic hypertension, acute coronary syndrome or cardiac surgery within the last 3 months.
5. Patients with known history or current treatment with cardiotoxic agents.
6. Receiving radiation on the left side of body.
7. History of rheumatic fever
8. Alcohol abuse.
9. Current participation in any other clinical investigation.
10. End-stage renal disease or patients on dialysis.
11. Patients with diabetic ketoacidosis or patients with type 1 diabetes mellitus.
12. Glomerular Filtration Rate <30ml/Kg/min.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
''Cardiac troponin T'' | Baseline and one time at the end of chemotherapy (3 to 5 days after the last dose of doxorubicin).
  Monitoring the serum biomarker Cardiac troponin T at baseline and one time at the end of chemotherapy after the last dose of doxorubicin.
  "The incidence of troponin elevation above the threshold indicated by the manufacturer of the assay used by the local laboratories will be recorded."
Echocardiography (ECHO) | Baseline, after each 3 doses of doxorubicin-based chemotherapy and 3 months after the end of chemotherapy.
  Initial evaluation of cardiac function guided by Echocardiography (ECHO) and clinical examination at baseline, after each 3 doses of doxorubicin-based chemotherapy and for follow up for 2 consecutive times every 3 months after the end of chemotherapy.
  "Cardiotoxicity or left ventricular dysfunction" will be defined as: a reduction of LV ejection fraction (LVEF) by 10% or more from baseline or with values lower than 50% at any follow up.

REFERENCES:
- [Result] Kaya MG, Ozkan M, Gunebakmaz O, Akkaya H, Kaya EG, Akpek M, Kalay N, Dikilitas M, Yarlioglues M, Karaca H, Berk V, Ardic I, Ergin A, Lam YY. Protective effects of nebivolol against anthracycline-induced cardiomyopathy: a randomized control study. Int J Cardiol. 2013 Sep 1;167(5):2306-10. doi: 10.1016/j.ijcard.2012.06.023. Epub 2012 Jun 22. PMID 22727976
- [Result] Janbabai G, Nabati M, Faghihinia M, Azizi S, Borhani S, Yazdani J. Effect of Enalapril on Preventing Anthracycline-Induced Cardiomyopathy. Cardiovasc Toxicol. 2017 Apr;17(2):130-139. doi: 10.1007/s12012-016-9365-z. PMID 27003392
- [Result] Broeyer FJ, Osanto S, Suzuki J, de Jongh F, van Slooten H, Tanis BC, Bruning T, Bax JJ, Ritsema van Eck HJ, de Kam ML, Cohen AF, Mituzhima Y, Burggraaf J. Evaluation of lecithinized human recombinant super oxide dismutase as cardioprotectant in anthracycline-treated breast cancer patients. Br J Clin Pharmacol. 2014 Nov;78(5):950-60. doi: 10.1111/bcp.12429. PMID 24844787
- [Result] Abuosa AM, Elshiekh AH, Qureshi K, Abrar MB, Kholeif MA, Kinsara AJ, Andejani A, Ahmed AH, Cleland JGF. Prophylactic use of carvedilol to prevent ventricular dysfunction in patients with cancer treated with doxorubicin. Indian Heart J. 2018 Dec;70 Suppl 3(Suppl 3):S96-S100. doi: 10.1016/j.ihj.2018.06.011. Epub 2018 Jun 18. PMID 30595329
- [Result] Kalay N, Basar E, Ozdogru I, Er O, Cetinkaya Y, Dogan A, Inanc T, Oguzhan A, Eryol NK, Topsakal R, Ergin A. Protective effects of carvedilol against anthracycline-induced cardiomyopathy. J Am Coll Cardiol. 2006 Dec 5;48(11):2258-62. doi: 10.1016/j.jacc.2006.07.052. Epub 2006 Nov 9. PMID 17161256
- [Result] Eliaa SG, Al-Karmalawy AA, Saleh RM, Elshal MF. Empagliflozin and Doxorubicin Synergistically Inhibit the Survival of Triple-Negative Breast Cancer Cells via Interfering with the mTOR Pathway and Inhibition of Calmodulin: In Vitro and Molecular Docking Studies. ACS Pharmacol Transl Sci. 2020 Nov 11;3(6):1330-1338. doi: 10.1021/acsptsci.0c00144. eCollection 2020 Dec 11. PMID 33344906
- [Result] Wang CY, Chen CC, Lin MH, Su HT, Ho MY, Yeh JK, Tsai ML, Hsieh IC, Wen MS. TLR9 Binding to Beclin 1 and Mitochondrial SIRT3 by a Sodium-Glucose Co-Transporter 2 Inhibitor Protects the Heart from Doxorubicin Toxicity. Biology (Basel). 2020 Oct 29;9(11):369. doi: 10.3390/biology9110369. PMID 33138323
- [Result] Baris VO, Dincsoy AB, Gedikli E, Zirh S, Muftuoglu S, Erdem A. Empagliflozin Significantly Prevents the Doxorubicin-induced Acute Cardiotoxicity via Non-antioxidant Pathways. Cardiovasc Toxicol. 2021 Sep;21(9):747-758. doi: 10.1007/s12012-021-09665-y. Epub 2021 Jun 5. PMID 34089496
- [Result] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A. Corrigendum to: 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure: Developed by the Task Force for the diagnosis and treatment of acute and chronic heart failure of the European Society of Cardiology (ESC) With the special contribution of the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2021 Dec 21;42(48):4901. doi: 10.1093/eurheartj/ehab670. No abstract available. PMID 34649282
- [Result] Sabatino J, De Rosa S, Tamme L, Iaconetti C, Sorrentino S, Polimeni A, Mignogna C, Amorosi A, Spaccarotella C, Yasuda M, Indolfi C. Empagliflozin prevents doxorubicin-induced myocardial dysfunction. Cardiovasc Diabetol. 2020 May 15;19(1):66. doi: 10.1186/s12933-020-01040-5. PMID 32414364
- [Result] Chang WT, Lin YW, Ho CH, Chen ZC, Liu PY, Shih JY. Dapagliflozin suppresses ER stress and protects doxorubicin-induced cardiotoxicity in breast cancer patients. Arch Toxicol. 2021 Feb;95(2):659-671. doi: 10.1007/s00204-020-02951-8. Epub 2020 Nov 19. PMID 33211168
- [Result] Oh CM, Cho S, Jang JY, Kim H, Chun S, Choi M, Park S, Ko YG. Cardioprotective Potential of an SGLT2 Inhibitor Against Doxorubicin-Induced Heart Failure. Korean Circ J. 2019 Dec;49(12):1183-1195. doi: 10.4070/kcj.2019.0180. Epub 2019 Jul 31. PMID 31456369
- [Result] Mustroph J, Wagemann O, Lucht CM, Trum M, Hammer KP, Sag CM, Lebek S, Tarnowski D, Reinders J, Perbellini F, Terracciano C, Schmid C, Schopka S, Hilker M, Zausig Y, Pabel S, Sossalla ST, Schweda F, Maier LS, Wagner S. Empagliflozin reduces Ca/calmodulin-dependent kinase II activity in isolated ventricular cardiomyocytes. ESC Heart Fail. 2018 Aug;5(4):642-648. doi: 10.1002/ehf2.12336. PMID 30117720
- [Result] Connelly KA, Zhang Y, Visram A, Advani A, Batchu SN, Desjardins JF, Thai K, Gilbert RE. Empagliflozin Improves Diastolic Function in a Nondiabetic Rodent Model of Heart Failure With Preserved Ejection Fraction. JACC Basic Transl Sci. 2019 Feb 25;4(1):27-37. doi: 10.1016/j.jacbts.2018.11.010. eCollection 2019 Feb. PMID 30847416
- [Result] Brzozowski JS, Skelding KA. The Multi-Functional Calcium/Calmodulin Stimulated Protein Kinase (CaMK) Family: Emerging Targets for Anti-Cancer Therapeutic Intervention. Pharmaceuticals (Basel). 2019 Jan 7;12(1):8. doi: 10.3390/ph12010008. PMID 30621060
- [Result] Cardinale D, Colombo A, Bacchiani G, Tedeschi I, Meroni CA, Veglia F, Civelli M, Lamantia G, Colombo N, Curigliano G, Fiorentini C, Cipolla CM. Early detection of anthracycline cardiotoxicity and improvement with heart failure therapy. Circulation. 2015 Jun 2;131(22):1981-8. doi: 10.1161/CIRCULATIONAHA.114.013777. Epub 2015 May 6. PMID 25948538